CLINICAL TRIAL: NCT06662838
Title: Evaluation of Ergonomics Awareness and First Aid Training Activities Given to Children of Seasonal Agricultural Worker Families
Brief Title: Ergonomics and First Aid Training for Children of Seasonal Agricultural Worker Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma BOZDAG, Associate Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HRU-BOZDAG-005
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Worker Disease, Agricultural
Keywords: child; ergonomics; first aid
MeSH Terms: conditions — Agricultural Workers' Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control grubu (No Intervention): Children will first be administered the Personal Information Form, Ergonomics Awareness Questionnaire for Children and First Aid Knowledge Level Questionnaire for Children. After one month without any intervention, Ergonomics Awareness Questionnaire for Children and First Aid Knowledge Level Questionnaire for Children will be administered to the children again.
- intervention group (Experimental): Children will first be administered the Personal Information Form, Ergonomics Awareness Questionnaire for Children and First Aid Knowledge Level Questionnaire for Children. Afterwards, children will be included in the Ergonomics Awareness and First Aid Training Program. One month after the training, Ergonomics Awareness Questionnaire for Children and First Aid Knowledge Level Questionnaire for Children will be administered again.
  Interventions: Other: Ergonomics Awareness and First Aid Training Program

INTERVENTIONS:
Other: Ergonomics Awareness and First Aid Training Program — The ergonomic awareness and first aid training program includes training on possible situations that children of seasonal agricultural worker families may encounter in the field.
  Arms: intervention group

SUMMARY:
The aim of this project is to evaluate the effectiveness of ergonomic awareness and first aid training given to children of seasonal agricultural worker families.

DETAILED DESCRIPTION:
In our country, especially from the Southeastern Anatolia region, the seasonal agricultural worker migration movement exceeding 1 million starts in March-April and ends in October-November. In Turkey, a significant number of children are forced to work in agriculture in more than 50 provinces in different regions of the country by participating in seasonal agricultural worker migration with their families. Şanlıurfa, which constitutes our project area, is the third largest agricultural area province in Turkey after Konya and Ankara. Despite this, due to reasons such as high population growth rate, mechanization in agriculture, division of agricultural lands by inheritance, and the failure of industry to develop in parallel with agricultural production, thousands of people migrate from Şanlıurfa to different regions of our country every year as seasonal migrant agricultural workers.

The "National Program to Combat Child Labor (2017-2023) Action Plan" was carried out by the Ministry of Labor and Social Security of the Republic of Turkey to eliminate child labor in our country. Similarly, among our 11th development goals (2019-2023), eliminating the worst forms of child labor in seasonal migratory agricultural work has been given priority. In this context, some projects such as the "Prevention of Child Labor in Seasonal Agriculture Project and the Comprehensive Model Project to Eliminate the Worst Forms of Child Labor in Seasonal Hazelnut Farming in Turkey" have been carried out in cooperation with the Ministry of Labor and Social Security, the International Labor Organization Turkey Office, labor and employer organizations, the Ministries of National Education, Interior, Agriculture and Forestry, the Turkish Employment Agency, municipalities, universities and non-governmental organizations in our country. These projects were generally carried out to identify and register MTİ children and ensure that they continue their education in the provinces they migrated to. The pilot provinces where these projects are carried out are generally provinces such as Şanlıurfa, Adıyaman, Mardin, Diyarbakır, where seasonal agricultural worker child migration is intense in our country, or Ordu, Sakarya, Malatya, Düzce, Adana, where seasonal agricultural worker children intensively go to work. However, many reasons such as earthquakes, pandemics and floods experienced in our country have prevented the desired goal from being achieved. In article 730 of our 12th development goals (2024-2028), priority has been given to continuing the fight against child labor with determination and providing first aid, occupational health and safety, children's rights and labor law training to seasonal migrant agricultural worker children. Şanlıurfa, where the project will be carried out, is among the provinces with the highest seasonal agricultural worker child migration in our country, and was affected by earthquake and flood in 2023 after the COVID-19 outbreak. It is also the 3rd province with the highest refugee population. The aim of this project is to evaluate the effectiveness of ergonomic awareness and first aid training given to children of seasonal agricultural worker families.

ELIGIBILITY:
Inclusion Criteria:

* Children who are between the ages of 14 and 18, who have no communication problems, who volunteer to participate in the research, and whose families have worked as seasonal agricultural workers at least once in their lives will be included in the study.

Exclusion Criteria:

* Children who do not meet the sample selection criteria, do not attend ergonomic awareness and first aid training, or drop out of training will be excluded from the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2024-12-08 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Ergonomics awareness level | 1 month
  Scores from the ergonomic awareness survey for children
First aid knowledge level | 1 month
  Scores from the first aid knowledge level survey for children

CONTACTS AND LOCATIONS:
Overall Officials: fatma bozdağ, Principal Investigator — Harran University
Locations (1):
- Fatma Bozdağ, Sanliurfa, Turkey (Türkiye)